CLINICAL TRIAL: NCT04600323
Title: Bicarbonate Administration and Cognitive Function in Midlife and Older Adults With CKD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-1672; R21AG068657 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Acidosis; Chronic Kidney Disease; Cognitive Dysfunction
MeSH Terms: conditions — Acidosis; Renal Insufficiency, Chronic; Cognitive Dysfunction | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo medication will be used at a dose of 0.5 mEq/kg-lean body weight/day
  Interventions: Drug: Placebo
- Sodium bicarbonate (Experimental): Sodium bicarbonate will be used at a dose of 0.5 mEq/kg-lean body weight/day.
  Interventions: Drug: Sodium Bicarbonate Tablets

INTERVENTIONS:
Drug: Sodium Bicarbonate Tablets — Participants will be given sodium bicarbonate at 0.5 mEq/kg-LBW/day for 12 months
  Arms: Sodium bicarbonate
Drug: Placebo — Participants will be given placebo at 0.5 mEq/kg-LBW/day for 12 months
  Arms: Placebo

SUMMARY:
This is a pilot, randomized, double-blinded, placebo-controlled, 12-month trial of 50 patients with CKD stage 3b-4 with metabolic acidosis to examine the effect of sodium bicarbonate therapy on cognitive and cerebrovascular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old
* Serum bicarbonate 16-22 mEq/L on 2 separate measurements (at least 1 day apart)
* CKD stage 3b or 4 at time of screening (eGFR 15-44 ml/min/1.73m2)
* Blood pressure <130/80 mm Hg prior to randomization
* Use of angiotensin converting enzyme inhibitor or angiotensin receptor blocker
* Stable anti-hypertensive regimen for at least one month prior to randomization
* Montreal Cognitive Assessment Score > 24
* No history of stroke
* No history of dementia
* No history of neurologic disease
* Able to provide consent

Exclusion Criteria:• Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year

* Use of chronic daily oral alkali within the last 3 months (including sodium bicarbonate, calcium carbonate or baking soda)
* Uncontrolled hypertension
* Serum potassium < 3.3 or ≥ 5.5 mEq/L at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known EF ≤30%, or hospital admission for heart failure within the past 3 months
* Factors judged to limit adherence to interventions
* Anticipated initiation of dialysis or kidney transplantation within 12 months
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Chronic use of supplemental oxygen

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.

REFERENCES:
- [Derived] Gu F, You Z, Hawkins N, Reddin R, Hamour R, Shapiro A, Coughlan C, Seals D, Furgeson S, Dixon A, Nowak KL, Kendrick J. Effects of sodium bicarbonate therapy on cognitive and cerebrovascular function in midlife and older adults with chronic kidney disease: a pilot randomized trial. BMC Nephrol. 2025 Aug 12;26(1):454. doi: 10.1186/s12882-025-04388-6. PMID 40797182
- [Derived] Perez L, You Z, Kendrick J. Association of Plant-Based Protein Intake with Cognitive Function in Adults with CKD. Kidney360. 2023 Nov 1;4(11):1554-1561. doi: 10.34067/KID.0000000000000278. Epub 2023 Oct 27. PMID 37889573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Sodium Bicarbonate
Started | 16 | 18
Completed | 16 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sodium Bicarbonate | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (5.9) | 62.0 (7.5) | 61.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34
Hypertension [Count of Participants; unit: Participants] | 16 | 16 | 32
Diabetes [Count of Participants; unit: Participants] | 10 | 12 | 22
Bicarbonate (mEq/L) [Mean (Standard Deviation); unit: mEq/L] | 21.8 (1.9) | 23.0 (1.5) | 22.7 (2.3)
GFR (ml/min/1.73m2) [Mean (Standard Deviation); unit: ml/min/1.73m2] | 32.8 (10.9) | 36.9 (16.7) | 34.8 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function Composite Score at 12 Months
Description: Cognitive function will be determined using the NIH Toolbox-Cognition Battery computerized tests. The Cognitive function composite score is based on the average of the Fluid and Crystallized composites. It is derived by averaging the Fluid and Crystallized standard scores, then deriving standard scores based on this new distribution. Fully Corrected T-scores are adjusted for for age, gender, race/ethnicity, and educational attainment. The score compares the score of the participant to those in the NIH Toolbox nationally representative normative sampling. The T-score has a mean of 50 in the general population and a SD of 10. Scores higher than the mean indicate better performance.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Sodium Bicarbonate
Number analyzed (Participants) | 16 | 17
T-score
  Baseline | 52.3 (8.8) | 47.3 (8.5)
  12 months | 53.5 (8.5) | 49.3 (11.0)

2. Primary Outcome: Change in Fluid Cognition Composite Score at 12 Months
Description: NIH Toolbox will be used to assess fluid cognition composite score. This score includes all the tests that are measuring fluid ability: Flanker, Dimensional Change, Picture sequence memory, list sorting and pattern comparison. The composite score is derived by averaging the standard scores of each of the measures. Fully Corrected T-scores are adjusted for age, gender, race/ethnicity, and educational attainment. The score compares the score of the participant to those in the NIH Toolbox nationally representative normative sampling. A fully corrected T-score at or near 50 (population mean with standard deviation of 10) indicates ability that is average compared with others nationally and one below 40 suggests the possibility of cognitive impairment. N
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Sodium Bicarbonate
Number analyzed (Participants) | 16 | 17
T-score
  Baseline | 52.1 (10.8) | 44.7 (8.7)
  12 months | 53.0 (9.4) | 46.9 (11.7)

3. Primary Outcome: Change in Crystallized Cognition Composite Score at 12 Months
Description: NIH Toolbox will be used to assess crystallized cognition composite score. This composite score includes the picture vocabulary and reading tests. The composite score is derived by averaging the standard scores of each of the measure, and then driving standard scores based on this new distribution. Fully Corrected T-scores are adjusted for age, gender, race/ethnicity, and educational attainment. The score compares the score of the participant to those in the NIH Toolbox nationally representative normative sampling. A fully corrected T-score at or near 50 (population mean with standard deviation of 10) indicates ability that is average compared with others nationally as the mean T-score is 50 nationally. A score higher than 50 indicates better crystallized cognition.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Sodium Bicarbonate
Number analyzed (Participants) | 16 | 17
T-score
  Baseline | 52.8 (8.3) | 49.6 (8.0)
  12 months | 53.5 (7.6) | 50.6 (9.0)

4. Secondary Outcome: Change in Cerebrovascular Reactivity at 12 Months
Description: Relative cerebrovascular reactivity was calculated as % change in mean blood flow velocity of the middle cerebral artery/(hypercapnia breath-by-breath end-tidal partial pressure of CO2 (ETCO2) minus resting ETCO2).
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent change/mmHg
Arm/Group | Placebo | Sodium Bicarbonate
Number analyzed (Participants) | 16 | 17
percent change/mmHg
  Baseline | 2.5 (1.4) | 2.4 (1.2)
  12 months | 2.7 (1.3) | 2.5 (1.1)

5. Secondary Outcome: Percent Change in Mean Blood Flow Velocity of the Middle Cerebral Artery at 12 Months
Description: Measured using Transcranial Doppler Ultrasonography in response to a vasodilatory hypercapnic challenge.The change in mean blood flow velocity of the middle cerebral artery (MVMCA) was computed as the difference between hypercapnic MVMCA and normocapnic MVMCA
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Sodium Bicarbonate
Number analyzed (Participants) | 16 | 17
percent change
  Baseline | 26.2 (17.0) | 22.6 (13.1)
  12 months | 32.3 (21.7) | 25.0 (12.4)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Sodium Bicarbonate
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/16 | 6/18
Other Adverse Events (participants affected / at risk) | 6/16 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Sodium Bicarbonate (N=18)
Hospitalization (Cardiac disorders) | 2 (2) | 3 (3)
Hospitalization (Infections and infestations) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Sodium Bicarbonate (N=18)
Dialysis initiation (Renal and urinary disorders) | 0 (0) | 2 (2)
New Lower Extremity Edema (Cardiac disorders) | 2 (2) | 3 (3)
Increase in antihypertensive therapy (Cardiac disorders) | 4 (4) | 4 (4)
Increase in diuretic therapy (Cardiac disorders) | 0 (0) | 3 (3)
High serum bicarbonate level (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT04600323/Prot_SAP_000.pdf